CLINICAL TRIAL: NCT02883595
Title: Efficacy of Thymosin Alpha 1 on Improving Monocyte Function for Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wu Jianfeng, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: thymosin alpha 1
Record Dates: First submitted 2016-08-10; First posted 2016-08-30 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Sepsis
Keywords: thymosin alpha 1; sepsis; monocyte; pharmacokinetics
MeSH Terms: conditions — Sepsis | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- thymosin alpha 1 (Experimental): Subcutaneous injections of 1.6 mg thymosin alpha 1 twice per day for seven days, the lyophilized powder is to be reconstituted with 1 ml of the provided diluent.
  Interventions: Drug: thymosin alpha 1
- Placebo (Placebo Comparator): Subcutaneous injections of placebo (saline) twice per day for seven days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: thymosin alpha 1 — Subcutaneous injections of 1.6 mg thymosin alpha 1 twice per day for seven days, prior to administration, the lyophilized powder is to be reconstituted with 1 ml of the provided diluent.
  Other Names: thymalfasin
  Arms: thymosin alpha 1
Other: Placebo — Subcutaneous injections of placebo (saline) twice per day for seven days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether thymosin alpha 1 is effective on improving monocyte function and has the desired pharmacologic activity for sepsis

DETAILED DESCRIPTION:
Part 1: To observe the function of thymosin alpha 1 in sepsis patients via improving phagocytosis, bacteria eradication and antigen-presenting on monocyte Part 2: Pharmacokinetics of thymosin alpha 1 for sepsis

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent from the patients or their next of kin for patients unable to consent
2. Age ≥18 yrs
3. Presence of sepsis/ septic shock according to sepsis 3.0

Exclusion Criteria:

1. Pregnant or lactation period.
2. Age <18 yrs
3. Receiving immunosuppressive therapy such as cyclosporine, azathioprine or cancer chemotherapy within one month.
4. History of bone marrow, lung, liver, kidney, pancreas or small bowel transplantation;
5. Acute pancreatitis with no established source of infection.
6. Not expected to survive 28 days because of end-stage diseases.
7. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Ta 1 improving immune function of monocyte for sepsis, used by flow cytometric to measure phagocytosis(CD11b, CD64), antigen presenting(HLA-DR, CD86 and PD-L1), and apoptosis(active caspase 3) on monocyte, | 28days
  Phagocytosis was measured by expression of monocyte surface antigen CD64 and CD11b, as well as pHrodo™ BioParticles® Phagocytosis Kits to assessing phagocytic activity on monocyte; antigen presenting was measured by HLA-DR, costimulatory molecule CD86 and inhibitory molecule PD-L1 on monocyte; apoptosis was measured by active caspase 3 on monocyte

SECONDARY OUTCOMES:
Relationship between concentration of Ta 1 and prognosis of sepsis patients, measured by concentration of Ta 1, 28-day all-cause mortality, 28-day clearance rate of pathogenic microorganism, ICU stays and hospital stays | 28 days
  Concentration of Ta 1 was measured on day 0, 3 and 7 after injection drug or placebo
Maximum observed serum concentration (Cmax) of Ta 1 | 7 days
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of Ta 1 | 7 days
Terminal serum half-life (T-HALF) of Ta 1 | 7 days
Time of maximum observed serum concentration (Tmax) of Ta 1 | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jianfeng, M. D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided